CLINICAL TRIAL: NCT02214615
Title: Pilot Study on the Response of Inherited Erythromelalgia Patients With NaV1.7 Mutations to Carbamazepine: Clinical Imaging Study
Brief Title: Carbamazapine for Inherited Erythromelalgia Patients With NaV1.7 Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SW0023
Record Dates: First submitted 2014-08-10; First posted 2014-08-12 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Erythromelalgia
MeSH Terms: conditions — Erythromelalgia | interventions — Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbamazepine (Active Comparator): Administered in gradual doses from 200 mg twice a day increasing to no more than 800 mg twice a day if symptoms do not reduce. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Interventions: Drug: Carbamazepine
- Placebo (Placebo Comparator): Administered in gradual doses from 200 mg twice a day increasing to no more than 800 mg twice a day if symptoms do not reduce to match dosing with carbamazepine. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbamazepine — Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day. Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
  Other Names: Tegretol
  Arms: Carbamazepine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This research study is designed to investigate brain response using fMRI scan, and behavioral responses, to treatment with the drug carbamazepine (CBZ) in patients with the painful sodium channelopathy inherited Erythromelalgia (IEM). This study is designed to identify the central nervous system (CNS) regions that are activated during ongoing or evoked pain attacks, and the altered CNS response to CBZ treatment. This will advance our understanding of how IEM affects the brain. We also hope to validate a pharmacogenic approach to the study of IEM by use of an FDA approved drug. We hope, but cannot be sure, that subjects will directly benefit from this study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis/symptoms of EM
* specific NaV1.7 sodium channel mutations (including S241T)

Exclusion Criteria:

* patients with no identified NaV1.7 mutation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Waxman, MD, PhD, Principal Investigator — VAMC West Haven and Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbamazepine Then Placebo: Administered in gradual doses from 200 mg twice a day increasing to no more than 800 mg twice a day if symptoms do not reduce. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Carbamazepine: Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day.
  Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
- Placebo Then Carbamazepine: Administered in gradual doses from 200 mg twice a day increasing to no more than 800 mg twice a day if symptoms do not reduce to match dosing with carbamazepine. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Placebo: Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day. Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
Period: First Intervention
Arm/Group | Carbamazepine Then Placebo | Placebo Then Carbamazepine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Washout
Arm/Group | Carbamazepine Then Placebo | Placebo Then Carbamazepine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Carbamazepine Then Placebo | Placebo Then Carbamazepine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Carbamazepine Then Placebo: Administered in gradual doses from 100 mg twice a day increasing to no more than 400 mg twice a day if symptoms do not reduce. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Carbamazepine: Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day.
  Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
- Placebo the Carbamazepine: Administered in gradual doses from 100 mg twice a day increasing to no more than 400 mg twice a day if symptoms do not reduce to match dosing with carbamazepine. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Placebo: Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day. Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
- Total: Total of all reporting groups
Arm/Group | Carbamazepine Then Placebo | Placebo the Carbamazepine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Erythromelalgia mutations S241T [Number; unit: participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Carbamazepine Affects Pain in Patients With S241T NaV1.7 IEM Mutation
Time Frame: 15 days
Measure: Number; unit: minutes
Arm/Group | Carbamazepine Then Placebo | Placebo Then Carbamazepine
Number analyzed (Participants) | 1 | 1
minutes
  Time in Pain Carbamazepine | 3015 | 136
  Time in Pain Placebo | 6360 | 915

2. Secondary Outcome: Carbamazepine Affects Mean Duration of Pain Episode
Time Frame: 15 days
Measure: Number; unit: minutes
Arm/Group | Carbamazepine Then Placebo | Placebo Then Carbamazepine
Number analyzed (Participants) | 1 | 1
minutes
  Mean episode duration with Carbamazepine | 274.1 | 45.3
  Mean episode duration with placebo | 615 | 91.5

ADVERSE EVENTS:
Groups:
- Carbamazepine: Administered in gradual doses from 100 mg twice a day increasing to no more than 400 mg twice a day if symptoms do not reduce. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Carbamazepine: Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day.
  Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
- Placebo: Administered in gradual doses from 100 mg twice a day increasing to no more than 400 mg twice a day if symptoms do not reduce to match dosing with carbamazepine. After 2 weeks of steady dose drug will be tapered down every 3 days.
  Placebo: Day 1: Take 200 mg twice a day. Day 2: Take 200 mg twice a day. Day 3: Take 200 mg twice a day. Day 4: Take 200 mg twice a day. Day 5: Take 400 mg twice a day. Day 6: Take 400 mg twice a day. Day 7: Take 400 mg twice a day. Day 8: Take 400 mg twice a day. Day 9: Take 600 mg twice a day. Day 10: Take 600 mg twice a day. Day 11: Take 600 mg twice a day. Day 12: Take 600 mg twice a day. Day 13: Take 800 mg capsules twice a day. Day 14: Take 800 mg twice a day. Day 15: 800 mg twice a day. Day 16: Take 800 mg twice a day.
  Taper Down (After Visit 4 and 7) If maximal dose of 800 mg/day has been achieved, tapering down will take 9 days Taper down for 600 mg/day will take 6 days, and for 400 mg/day will take 3 days.
Arm/Group | Carbamazepine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
all subjects had to have erythromelalgia SCN9A mutation S241T

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No